CLINICAL TRIAL: NCT00459810
Title: A Phase II Study of Paclitaxel Poliglumex (PPX) in Combination With Transdermal Estradiol for the Treatment of Androgen Independent Prostate Cancer After Docetaxel Chemotherapy
Brief Title: Paclitaxel Poliglumex and Estradiol in Treating Patients With Stage IV Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540438; OHSU-2656 (Other: OHSU IRB)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — paclitaxel poliglumex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: transdermal estradiol — Transdermal estradiol given 0.2mg/day for duration of study.
Drug: paclitaxel poliglumex — Paclitaxel poliglumex (PPX) is a macromolecular polymer-drug conjugate of paclitaxel. PPX was given every 28 days, at a dose of 150 mg/m2

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel poliglumex, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Estradiol may kill prostate cancer cells that no longer respond to hormone therapy. Giving paclitaxel poliglumex together with estradiol may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel poliglumex together with estradiol works in treating patients with stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the PSA response rate in patients with androgen independent metastatic prostate cancer treated with paclitaxel poliglumex and transdermal estradiol.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the response rate in patients treated with this regimen.
* Determine the time to PSA progression and measurable disease progression in patients treated with this regimen.
* Determine time to death from all causes in patients treated with this regimen.
* Correlate levels of serum estradiol, serum cathepsin B, and bone turnover markers with PSA response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive transdermal estradiol continuously (patches changed every 7 days) until the PSA level rises. Patients whose PSA increases above baseline or PSA decreases < 10% after 4 weeks of estradiol therapy or whose serum PSA reduction is < 50% after 12 weeks of estradiol therapy also receive paclitaxel poliglumex therapy. These patients receive paclitaxel poliglumex IV over 10-20 minutes on day 1. Treatment with paclitaxel poliglumex repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Stage IV disease

    * Radiographic evidence of regional or distant metastases
* Evidence of disease progression (by PSA and/or imaging studies) despite standard hormonal therapy and after exposure to docetaxel-containing chemotherapy, as evidenced by any of the following:

  * Measurable or evaluable disease progression, defined as the appearance of new lesion(s) or unequivocal increase in previously existing lesions or masses
  * Disease progression by PSA*, defined by 1 of the following:

    * 3 consecutively rising PSA with the second PSA taken ≥ 1 week after the first PSA
    * 2 consecutively rising PSA with a fourth PSA > the second PSA NOTE: *The last required PSA must be after the required antiandrogen washout period for patients who have been on antiandrogen therapy
* Must have received prior therapy with at least two 3-weekly doses or six weekly doses of docetaxel

  * Patients may have discontinued therapy due to progression, intolerance, completion of planned therapy, or other reasons
  * Prior treatment with combinations of docetaxel with estramustine phosphate sodium or noncytotoxic agents (biologic agents) allowed
* Serum testosterone < 50 ng/dL (unless surgically castrate)

  * Patients must continue androgen deprivation with a luteinizing hormone-releasing hormone agonist if they have not undergone orchiectomy
* No known or suspected brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* No other active malignancy except adequately treated nonmelanoma skin cancer or other noninvasive or in situ neoplasm
* No other significant active medical illness or infection that would preclude study compliance
* No significant cardiovascular illness, including any of the following:

  * NYHA class III or IV congestive heart failure
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Acute deep venous thrombosis
  * Acute pulmonary embolism
* No significant peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior antiandrogen therapy (4 weeks for flutamide)

  * No current evidence of an antiandrogen withdrawal response
* More than 4 weeks since prior radiotherapy
* More than 8 weeks since prior radiopharmaceutical therapy (strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium)
* No prior paclitaxel
* No other concurrent cytotoxic agents
* No other concurrent chemotherapy or biologic response modifiers
* No concurrent supplements known or suspected to contain supplemental estrogens

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - OHSU Knight Cancer Institute, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-one patients enrolled in the trial between March 2007 and May 2008 in the medical clinics at Oregon Health & Science University and the University of California at San Francisco.
Groups:
- Transdermal Estradiol and Paclitaxel Poliglumex: All subjects enrolled were treated with transdermal estradiol 0.2 mg/24 hours for 4 weeks followed by the same dose of transdermal estradiol and paclitaxel poliglumex PPX 150 mg/m2 IV every 28 days.
Period: Overall Study
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response Rate: Number of Subjects With Decreases in PSA of at Least 50%
Description: PSA response rate is defined at the number of patients who experienced a PSA decline of equal to or greater than 50%, confirmed by a second measurement at least 4 weeks later.
Time Frame: While receiving study agents (on average, 3 months)
Measure: Number; unit: Participants
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: Measurable Disease Response Rate (Soft Tissue)
Description: Measurable disease response rate by RECIST criteria. Response is defined as at least a 30% decrease in the sum of the longest diameter in measurable lesions (larger than 10mm at baseline).
Time Frame: While receiving study agents (on average, 3 months)
Measure: Number; unit: Participants
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Number analyzed (Participants) | 21
Participants | 0

3. Secondary Outcome: Time to Disease Progression
Description: Time from Day 1 to Day of meeting criteria for PSA or Measurable Disease Progression
Time Frame: At time of progression by PSA or RECIST criteria
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Number analyzed (Participants) | 21
Days | 28 [26 to 30]

4. Secondary Outcome: Time to Death
Description: Defined as time from Day 1 of study regimen to Date of death from any cause.
Time Frame: Measured at Date of Death from any cause
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Number analyzed (Participants) | 21
Months | 7.8 [4.8 to 10.8]

5. Secondary Outcome: Correlation of Levels of Serum Estradiol, Serum Cathepsin B, and Bone Turnover Markers With PSA Response
Description: These correlative analyses were not completed. As there were no PSA responses, it was not possible to correlate serum estradiol, serum cathepsin B, or bone turnover markers with PSA response.
Time Frame: Measured after 4 cycles of combination therapy
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: While on study agents
Arm/Group | Transdermal Estradiol and Paclitaxel Poliglumex
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol and Paclitaxel Poliglumex (N=21)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) — Subject admitted for gastric hemorrhage and thrombocytopenia. Event determined to be possibly related to study agents.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject admitted with lethargy, cough and elevated temperature. Chest X-ray demonstrated pneumonitis. Event determined to be possibly related to study agents.
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) — Subject admitted for intractable nausea and vomiting. Abdominal ultrasound was normal. Event deemed possibly related to study agents
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol and Paclitaxel Poliglumex (N=21)
hemoglobin decreased (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 3 (20)
Lymphopenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 3
Anorexia (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 7
Edema (Blood and lymphatic system disorders) | 2
Alkaline Phosphatase increased (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 11
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Breast pain (Reproductive system and breast disorders) | 4
Gynecomastia (Reproductive system and breast disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days